CLINICAL TRIAL: NCT03441516
Title: Effect of Choline Alphoscerate on Cognitive Function in Alzheimer's Dementia: A Multi-center, Randomized, Open-label, Pilot Study
Brief Title: Effect of Choline Alphoscerate on Cognitive Function in Alzheimer's Dementia
Acronym: ALFO-AD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YMC034
Record Dates: First submitted 2018-02-05; First posted 2018-02-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alfoatirin® Tab. + Aripezil® Tab. (Experimental): Choline Alphoscerate 400mg bid + Donepezil 10mg qd for 24 weeks
  Interventions: Drug: Alfoatirin® Tab. + Aripezil® Tab.
- Aripezil® Tab. (Active Comparator): Donepezil 10mg qd for 24 weeks
  Interventions: Drug: Aripezil® Tab.

INTERVENTIONS:
Drug: Alfoatirin® Tab. + Aripezil® Tab. — Choline Alphoscerate 400 mg Oral Tablet bid + Donepezil 10 mg Oral Tablet qd for 24 weeks
  Arms: Alfoatirin® Tab. + Aripezil® Tab.
Drug: Aripezil® Tab. — Donepezil 10 mg Oral Tablet qd for 24 weeks
  Arms: Aripezil® Tab.

SUMMARY:
This study will evaluate the performance of Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog) in patients with Alzheimer's disease (AD).

ELIGIBILITY:
Inclusion Criteria:

* 50 - 90 years of age
* Clinical diagnosis of dementia of the Alzheimer type determined by Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria
* A diagnosis of probable Alzheimer's Disease, or mild to moderate AD determined by NIA-AA (National Institute on Aging and the Alzheimer's Association) criteria
* K-MMSE score of 12 - 26
* Global Clinical Dementia Rating (CDR) score of 0.5 - 2
* Patient taking 10 mg of donepezil per day for a minimum of 12 weeks with a stable dose, not taking other brain pills including choline alfoscerate for at least 2 weeks from screening. Drugs that are likely to affect cognition are permissible if the dose is regular and stable for at least 2 weeks before screening and if the treatment continues for the duration of the trial.

Exclusion Criteria:

* Subject suspected of dementia due to organic causes other than Alzheimer's type dementia
* Other degenerative brain diseases or major mental illnesses such as major depression, bipolar disorder, alcohol/substance abuse or dependence, delirium
* Hypersensitive to choline alfoscerate, donepezil hydrochloride, or piperidine derivatives or the components of this drug
* Subject who has contraindications as listed in the SPC of choline alfoscerate or donepezil hydrochloride
* Other than the above who is deemed to be ineligible to participate in the trial

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
ADAS-cog | At 24 weeks
  To evaluate cognitive function

SECONDARY OUTCOMES:
ADAS-cog | At 12 weeks
  To evaluate cognitive function
K-MMSE (Korean version of Mini-Mental State Examination) | At 12 and 24 weeks
  To evaluate cognitive function
FAB (Frontal Assessment Battery) | At 12 and 24 weeks
  To evaluate frontal lobe dysfunction
S-IADL (Seoul-Instrumental Activities of Daily Living) | At 12 and 24 weeks
  To evaluate daily activities of living
CGA-NPI (Caregiver-Administered Neuropsychiatric Inventory) | At 12 and 24 weeks
  To evaluate neuropsychiatric symptom in dementia
Changes in brain metabolism by F-18 FDG brain PET | At 24 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - Dong-A University Hospital, Busan
  - Gyeongsang National University Hospital, Busan
  - Inje University Busan Paik Hospital, Busan
  - Inje University Haeundae Paik Hospital, Busan
  - Pusan National University Yangsan Hospital, Busan
  - Samsung Changwon Hospital, Busan